CLINICAL TRIAL: NCT01125111
Title: The Clinical Study of Making the Evidence With Application of Da Vinci-Robot Assisted Low Anterior Resection in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Nam Kyu Kim/Professor, Yonsei University, College of Medicine
Other Study IDs: 4-2009-0210
Record Dates: First submitted 2010-05-10; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- robotic surgery group
  Interventions: Procedure: surgery(robot versus laparoscopy)
- laparoscopic surgery group
  Interventions: Procedure: surgery(robot versus laparoscopy)

INTERVENTIONS:
Procedure: surgery(robot versus laparoscopy)

SUMMARY:
The clinical study of making the evidence with application of Da vinci-Robot assisted low anterior resection in rectal cancer

ELIGIBILITY:
Inclusion Criteria:

* 75 > age > 20
* Rectal cancer
* Non-distance metastasis
* Agree with this study

Exclusion Criteria:

* Benign prostate hyperplasia
* Previous history of urinary bladder or prostate gland operation
* Severe erectile dysfunction
* Defined as patients whose erectile scores were less than 10 in a preoperative questionnaire of the International Index of Erectile Function (IIEF)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who visit Severance Hospital for rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The difference in 1 month between two surgical methods in terms of Bladder function. | 1 month
  The robotic surgery for rectal cancer seemed to be associated with a much earlier recovery of normal voiding and sexual function compared to those of laparoscopic surgery although it needs to be verified by larger prospective comparative studies

SECONDARY OUTCOMES:
The difference in 3 months between two surgical methods in tems of Sexual function. | 3 months
The serial change of Bladder and sexual function according to times, in each operation method.

CONTACTS AND LOCATIONS:
Overall Officials: Nam Kyu Kim, Principal Investigator — Department of Surgery, Yonsei University College of Medicine, Seoul, Korea